CLINICAL TRIAL: NCT01817270
Title: A Study to Evaluate the Immunogenicity and Safety of 2 Doses of Live Attenuated Varicella Vaccine
Brief Title: Immunogenicity and Safety Study of 2 Doses of Live Attenuated Varicella Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changchun Keygen Biological Products Co., Ltd. (Other)
Collaborators: Guangdong Provincial Institute of Biological Products And Materia Medica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCT02038506
Record Dates: First submitted 2013-03-04; First posted 2013-03-25 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Chickenpox
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Live Attenuated Varicella Vaccine (Experimental): use the left arm flank deltoid muscle adheres to stick cohere place the skin after 75% ethyl alcohol disinfection the hypodermic injection
  Interventions: Biological: Live Attenuated Varicella Vaccine

INTERVENTIONS:
Biological: Live Attenuated Varicella Vaccine

SUMMARY:
The purpose of this study is to observe the occurrence of adverse events, seroconversion rate and geometric mean titres(GMTs) of 2 doses of live attenuated varicella vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal acceptable representative is willing and able to understand the protocol requirements and provide informed consent
* Participant is aged ≥ 1 year to ≤ 3 years
* Participant without preventive inoculation of varicella vaccine and previous history of chickenpox and zoster
* Subject and parent/guardian able to attend all scheduled visits and comply with all trial procedures
* Body temperature ≤ 37.5℃

Exclusion Criteria:

* Known allergy to any constituent of the vaccine
* Known acute illness, severe chronic disease, acute exacerbation of chronic disease and fever
* Known or suspected impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin since birth
* Reported the history of allergies, convulsions, epilepsy, mental illness and brain disease and clear serious systemic reaction
* Failed to the Expanded Programme on Immunization(EPI)
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination
* Plan to receive any vaccine in the 4 weeks following the trial vaccination
* Known bleeding disorder
* Receipt of whole blood, blood plasma or immunoglobulin in the 5 months preceding the trial vaccination
* Reported the history of acute illness had need systemic antibiotics or anti-viral treatment of infections in the 7 days preceding the trial vaccination
* An acute illness with or without fever (temperature ≥ 38.0℃) in the 3 days preceding enrollment in the trial
* Participation in any other interventional clinical trial
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the vaccine

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 368 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate and GMTs for live attenuated varicella vaccine | 35-42 days after the first and second doses

SECONDARY OUTCOMES:
Occurrence of adverse events | within 30 days after each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Huizhen Zheng, Master, Principal Investigator — Guangdong Center for Disease Prevention and Control
Locations (1):
- Xinxing Center for Disease Control and Prevention, Yunfu, Guangdong, China